CLINICAL TRIAL: NCT01122069
Title: Contrast Echocardiography in Assessment of Myocardial Perfusion in Patients With Non-ST Elevation Myocardial Infarction
Brief Title: Contrast Echocardiography in Non-ST Elevation Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: University of Bergen (Other)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Eva Gerdts, Professor of Cardiology, University of Bergen
Other Study IDs: MCE-NSTEMI; REK237.07 (Other: Regional Ethics Committee West Norway)
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Non-ST-Elevation Myocardial Infarction
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction | interventions — perflutren

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Contrast echocardiography: 110 patients with acute non-ST elevation myocardial infarct were examined with contrast echocardiography prior to coronary angiography.
  Interventions: Other: Perflutren Lipid Microsphere ultrasound contrast

INTERVENTIONS:
Other: Perflutren Lipid Microsphere ultrasound contrast — Perflutren Lipid Microsphere ultrasound contrast 0.01 ml/kg administered as intravenous bolus
  Other Names: Luminity

SUMMARY:
In patients with acute myocardial infarction, treatment logistics are primarily defined based upon ST segment shift in the electrocardiogram. While patients with ST elevation (STEMI) are forwarded to immediate coronary angiography and percutaneous coronary intervention, patients without ST elevation (NSTEMI) are initially medically treated and recommended coronary angiography within 48-72 hours.

Early invasive treatment has been found cost-effective in intermediate and high-risk NSTEMI patients and current guidelines recommend use of the Thrombolysis in Myocardial Infarction (TIMI) risk score to identify patients who will benefit from early intervention due to high risk of new infraction and cardiovascular death. However, new research has suggested that TIMI risk score may not always identify patients with severe angiographic disease.

The purpose of this study was to assess if contrast echocardiography could be used to identify NSTEMI patients with angiographically severe disease independent of their TIMI risk score.

ELIGIBILITY:
Inclusion Criteria:

* acute non-ST elevation myocardial infarction

Exclusion Criteria:

* hemodynamic unstable
* mechanical prosthetic heart valve
* severly reduced pulmonary function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 110 patients with acute non-ST elevation myocardial infarction
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2008-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mai Tone Lønnebakken, MD, Principal Investigator — University of Bergen, Bergen, Norway
Locations (1):
- Department of Heart Disease, Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Derived] Eskerud I, Gerdts E, Nordrehaug JE, Lonnebakken MT. Global Coronary Artery Plaque Area is Associated with Myocardial Hypoperfusion in Women with Non-ST Elevation Myocardial Infarction. J Womens Health (Larchmt). 2015 May;24(5):367-73. doi: 10.1089/jwh.2014.4920. Epub 2015 Feb 18. PMID 25692527
- [Derived] Lonnebakken MT, Nordrehaug JE, Gerdts E. No gender difference in the extent of myocardial ischemia in non-ST elevation myocardial infarction. Eur J Prev Cardiol. 2014 Jan;21(1):123-9. doi: 10.1177/2047487312454107. Epub 2012 Jul 2. PMID 22752464